CLINICAL TRIAL: NCT06600256
Title: Viz HCM (ECG Assist) Utilization Workflow Pilot
Status: Completed | Type: Observational
Sponsor: Viz.ai, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Viz-HCM-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pre-Viz: The number of HCM diagnosed patients (based on hospital records over the 6 months prior to site activation with the Viz HCM software) [pre-Viz]
  Interventions: Behavioral: Baseline Effectiveness Cohort
- post-Viz: The number of HCM patients (flagged by Viz HCM and confirmed by follow-up transthoracic ECHO and/or CMR diagnostic imaging) after site activation with the Viz HCM software [post-Viz]
  Interventions: Behavioral: Viz HCM ECG Review

INTERVENTIONS:
Behavioral: Viz HCM ECG Review — Viz HCM will auto-alert relevant users to ECGs the algorithm has deemed as suspicious for HCM. Following review of this alert and the patient's Medical/Clinical History, the reviewer will take the next Standard of Care action they deem appropriate.
  Groups: post-Viz
Behavioral: Baseline Effectiveness Cohort — A review of the timing and clinical details of the diagnostic process for patients diagnosed with HCM before the site began using Viz HCM.
  Groups: pre-Viz

SUMMARY:
This is a prospective, open-label, multi-center workflow pilot. Viz HCM will be implemented at each participating site and all conforming incoming ECG recordings within a 6-month enrollment period will be analyzed using Viz HCM. This workflow pilot provides an opportunity to understand how Viz HCM will be utilized and adopted post-market and to learn the pre- versus post-implementation impact of Viz HCM on HCM clinical workflow.

This pilot is designed to evaluate the implementation of Viz HCM for use in traditional HCM clinical workflow. Findings from this pilot will help inform the following:

* The impact of Viz HCM on HCM clinical workflow
* How Viz HCM will be utilized and adopted post-market
* The diversity in the HCM patient population and the variation in HCM clinical workflow

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a genetic cardiac disease that causes the walls of the lower heart chambers to thicken and stiffen. As the disease progresses, thickened walls around the left ventricle may block or reduce blood flow to the aorta, potentially interrupting the flow of oxygenated blood to the rest of the body. As a result, the heart must pump harder to overcome this obstruction and supply the body's circulation. HCM is initially suspected by the presence of an abnormal electrocardiogram (ECG) and confirmed by diagnostic imaging showing a left ventricular wall thickness of >15mm (>13mm in relatives of individuals with HCM or those who are genotype positive) that cannot be explained by another cardiac or general disease. The prevalence of HCM in the general population is 1:200 to 1:500 (~750,000 Americans); however only 10-20% of cases are diagnosed, signifying an under-recognition of HCM in clinical practice and thus a need for better disease detection.

Viz HCM is a software device designed to alert and triage suspected HCM patients to the appropriate clinical care team. The device consists of an artificial intelligence algorithm embedded in a standalone mobile application. This is a prospective, open-label, multi-center workflow pilot. Viz HCM will be implemented at each participating site and all conforming incoming ECG recordings within a 6-month enrollment period will be analyzed using Viz HCM. The pilot will measure device utilization based on the percentage of HCM suspected notifications viewed by users. Among the number of viewed Viz suspected HCM cases, data will also be collected on time to follow-up as well as the type, date, and number of follow-up tests after notification. Impact of Viz HCM on clinical workflow will be established by comparing the number of HCM diagnosed patients (based on hospital records over the 6 months prior to site activation) [pre-Viz] to the number of HCM patients (flagged by Viz HCM and confirmed by follow-up transthoracic ECHO and/or CMR diagnostic imaging) after site activation [post-Viz]

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of greater at the time of arrival to healthcare facility
* Patients underwent resting 12-lead digital electrocardiogram (ECG) at healthcare facility

Exclusion Criteria:

* Patients with poor or incomplete recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the 6-month enrollment period, patients who receive an ECG at participating sites will be screened to determine if they meet eligibility criteria. All patients meeting eligibility criteria will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Viz suspected HCM cases viewed by users | up to 10 minutes
  Algorithm performance - sensitivity and specificity of the Viz HCM software
Number of viewed Viz suspected HCM cases that receive any follow-up action (e.g., schedule test, physician referral) | up to 10 minutes
  algorithm processing time

SECONDARY OUTCOMES:
Number of HCM diagnosed patients (based on hospital records over the 6 months prior to site activation) [pre-Viz] | up to 10 minutes
  algorithm sensitivity
Number of HCM patients (flagged by Viz HCM and confirmed by follow-up transthoracic ECHO and/or CMR diagnostic imaging) [post-Viz] | up to 10 minutes
  algorithm specificity

OTHER OUTCOMES:
Type, date, and number of follow-up tests after HCM notification | 180 days
  exploratory endpoint
Time from HCM notification view to follow-up testing and/or documented diagnosis | up to 48 hours
  exploratory endpoint
User satisfaction (Viz HCM Physician Satisfaction Survey) | 180 days
  exploratory endpoint
Descriptive statistics by site and by patient demographic breakdown (e.g., race/ethnicity) | 180 days
  exploratory endpoint

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UC San Diego Sulpizio Cardiovascular Center, La Jolla, California
  - The Valley Hospital, Ridgewood, New Jersey
  - The Mount Sinai Hospital, New York, New York
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - HCA Methodist, San Antonio, Texas